CLINICAL TRIAL: NCT07090694
Title: Transcrestal Sinus Elevation With or Without PRF for Atrophic Maxilla: A Randomized Clinical Evaluation
Brief Title: PRF vs. Graftless Sinus Lift With Implant Placement
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Dar Al Uloom University (Other)
Responsible Party: Principal Investigator, Sally Abd-ElMeniem ElHaddad, Assist. Prof. Periodontology and Oral Medicine, Dar Al Uloom University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 038- 003- 2025
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Maxillary Sinus Floor Augmentation; Alveolar Bone Loss; Atrophy; Platelet-rich Fibrin; Dental Implant
Keywords: Transcrestal Sinus Lift; Crestal Approach Sinus Floor Elevation; Maxillary Sinus Augmentation; Platelet-Rich Fibrin; Single-Stage Implant Placement; Atrophic Posterior Maxilla
MeSH Terms: conditions — Alveolar Bone Loss; Atrophy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graftless Sinus Elevation with Simultaneous Implant Placement (Experimental): Participants in this arm undergo crestal sinus floor elevation without the use of any grafting material. The procedure involves a transcrestal (internal) sinus lift through sequential osteotomy followed by immediate placement of dental implants. The elevated sinus membrane is maintained by the implant fixture alone, allowing for natural blood clot formation and spontaneous bone regeneration.
  Interventions: Procedure: Graftless Transcrestal Sinus Floor Elevation with Immediate Implant Placement
- PRF-Grafted Sinus Elevation with Simultaneous Implant Placement (Active Comparator): Participants in this arm undergo crestal sinus floor elevation using platelet-rich fibrin (PRF) as the sole grafting material. PRF is prepared from the patient's own blood via centrifugation and inserted into the osteotomy site. A dental implant is then placed immediately, supporting the sinus membrane and serving as a tent for guided bone regeneration. This technique utilizes PRF's growth factors to promote healing and enhance new bone formation beneath the elevated sinus membrane.
  Interventions: Biological: Platelet-Rich Fibrin (PRF)-Assisted Transcrestal Sinus Floor Elevation with Immediate Implant Placement

INTERVENTIONS:
Procedure: Graftless Transcrestal Sinus Floor Elevation with Immediate Implant Placement — This intervention involves a minimally invasive internal (crestal) sinus lift performed without the use of any grafting material. The sinus membrane is elevated using sequential osteotomy drills, and a dental implant is immediately placed into the prepared site. The implant fixture acts as a tent pole, maintaining the lifted membrane and allowing for spontaneous bone regeneration through blood clot formation alone. This graftless method eliminates the need for additional biomaterials and is intended for patients with residual alveolar bone height of 5-7 mm
  Arms: Graftless Sinus Elevation with Simultaneous Implant Placement
Biological: Platelet-Rich Fibrin (PRF)-Assisted Transcrestal Sinus Floor Elevation with Immediate Implant Placement — This intervention utilizes autologous platelet-rich fibrin (PRF) as the sole grafting material during transcrestal sinus floor elevation. PRF is prepared from the patient's own venous blood using centrifugation and inserted into the osteotomy site after sinus membrane elevation. A dental implant is placed simultaneously to support the sinus membrane and stabilize the graft. The biologically active PRF matrix provides a scaffold rich in growth factors (e.g., TGF-β, PDGF, VEGF), promoting accelerated healing and enhanced bone formation beneath the elevated sinus floor. This technique is performed in a single-stage procedure, eliminating the need for synthetic or allogeneic grafts.
  Arms: PRF-Grafted Sinus Elevation with Simultaneous Implant Placement

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of sinus floor elevation using platelet-rich fibrin (PRF) compared to a graftless approach in adult patients with atrophic posterior maxilla (residual bone height 5-7 mm) requiring dental implant rehabilitation. The main questions it aims to answer are:

Does PRF enhance bone height gain more effectively than graftless sinus elevation? Does PRF improve implant stability and reduce marginal bone loss compared to the graftless approach? Researchers will compare the outcomes of PRF-grafted implants versus non-grafted implants to see if PRF improves radiographic and clinical results in single-stage implant placement.

Participants will:

Undergo internal sinus lift via crestal drilling approach

Be randomly assigned to one of two groups:

Group I: sinus lift without graft material Group II: sinus lift with PRF as the sole grafting material Receive simultaneous dental implant placement during the sinus lift Be monitored through clinical exams and radiographic imaging over 6 months postoperatively

DETAILED DESCRIPTION:
This randomized controlled clinical trial investigates the clinical and radiographic outcomes of crestal sinus floor elevation in the atrophic posterior maxilla, comparing two approaches: one using platelet-rich fibrin (PRF) as a sole grafting material and another performed without any grafting material. Both interventions are combined with single-stage dental implant placement. The rationale for this study is based on emerging evidence suggesting that graftless techniques, relying on blood clot stabilization and tenting of the sinus membrane, may be sufficient to induce predictable bone formation, especially when residual alveolar bone height is ≥5 mm.

The study involves adult patients presenting with edentulous posterior maxillary regions and limited vertical bone height due to sinus pneumatization and ridge resorption.

Participants are randomly allocated to either PRF or graftless groups. Both groups undergo transcrestal sinus elevation through sequential osteotomy, followed by immediate implant placement under a standardized surgical and prosthetic protocol.

Primary outcomes include radiographic bone gain and implant stability quotient (ISQ), while secondary outcomes include marginal bone loss and peri-implant clinical parameters. Radiographic evaluation is conducted using CBCT imaging at baseline and 6 months postoperatively. This study aims to provide evidence on whether PRF offers added clinical benefit over natural healing and clot formation in sinus lift procedures performed via the less invasive crestal approach.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 25 to 65 years
* Patients with one or more missing posterior maxillary teeth
* Residual alveolar bone height between 5 mm and 7 mm, confirmed by CBCT
* Good oral hygiene and motivation for implant therapy
* Adequate inter-arch space for prosthetic rehabilitation
* Absence of maxillary sinus pathology on radiographic assessment
* Patients willing to undergo single-stage implant placement with sinus lift
* Signed informed consent

Exclusion Criteria:

* Systemic diseases or medical conditions affecting bone metabolism or wound healing (e.g., uncontrolled diabetes, osteoporosis, immunocompromised status)
* History of radiation therapy in the head and neck region
* Use of medications influencing bone turnover (e.g., bisphosphonates, corticosteroids)
* Active periodontal disease or poor oral hygiene
* Smoking or tobacco use
* Parafunctional habits such as bruxism or clenching
* Pregnancy or breastfeeding
* Known bleeding disorders or abnormal coagulation profiles
* Presence of maxillary sinus infection or pathology
* Inability to attend follow-up visits or comply with study protocol

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Radiographic Bone Height Gain | Baseline and 6 months postoperatively
  Vertical bone gain measured using Cone Beam Computed Tomography (CBCT) from the alveolar crest to the elevated sinus floor. The measurement is taken at baseline (preoperatively) and compared with measurements at 6 months postoperatively to evaluate the success of sinus augmentation.

SECONDARY OUTCOMES:
Implant Stability Quotient (ISQ) | Immediate postoperative (Day 0) and 6 months postoperatively
  Measurement of primary and secondary implant stability using an Osstell device. ISQ values are recorded at the time of implant placement and at 6 months postoperatively to assess osseointegration and mechanical stability.
Marginal Bone Loss | Baseline and 6 months postoperatively
  Radiographic evaluation of crestal bone loss measured at the mesial and distal aspects of the implant using CBCT or standardized periapical radiographs. The difference in marginal bone height from baseline to 6 months will be calculated to assess peri-implant bone preservation.

CONTACTS AND LOCATIONS:
Overall Officials: SREIC College of Dentistry, Dar AlUloom University, Scientific Committee, Study Director — Dar AlUloom University, SA
Locations (1):
- College of Dentistry, Dar AlUloom University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Demographic data (age, sex)
  Baseline clinical measurements (residual bone height, CBCT parameters)
  Implant stability quotient (ISQ) values
  Radiographic bone gain and marginal bone loss measurements
  Adverse events or complications (if any)
Supporting Information: Study Protocol
Time Frame: IPD will be available within 6 months after publication of the primary study results, and for 6 month Data will be shared upon reasonable request through direct communication with the principal investigator. Access may be granted via secure data transfer or institutional repository, subject to data use agreement.
Access Criteria: Qualified researchers affiliated with academic institutions or regulatory bodies for non-commercial purposes.